CLINICAL TRIAL: NCT01123889
Title: Treatment of Rotator Cuff Syndrome With Injection of Autologous Platelet Rich Plasma
Brief Title: Treatment of the Rotator Cuff Disease With Platelet Rich Plasma Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Montri D. Wongworawat, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59322
Record Dates: First submitted 2010-04-20; First posted 2010-05-14 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Subacromial Impingement Syndrome; Partial Thickness Rotator Cuff Tear
Keywords: subacromial impingement; partial thickness rotator cuff; PRP; platelet rich plasma
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Ropivacaine; Lidocaine; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): corticosteroid injection into subacromial space
  Interventions: Drug: corticosteroid injection
- experimental (Experimental): patients will receive an injection of platelet rich plasma into the subacromial space
  Interventions: Biological: platelet rich plasma injection

INTERVENTIONS:
Biological: platelet rich plasma injection — 45 ml of a patient's own blood will be collected via blood draw, maintaining sterile technique. This will then be spun down using a Magellan Autologous Platelet Separator System, yielding platelet rich plasma (PRP). Under sterile conditions, patients will receive a 5 cc PRP injection (consisting of their own PRP) with 1 cc of 1% lidocaine and 1 cc of 0.5% ropivacaine into the subacromial space, administered by an orthopedic surgeon. This will be done using a posterior lateral approach. The patient will be monitored for 10 minutes in clinic for adverse reactions.
  Other Names: platelet rich plasma - PRP; naropin; xylocaine
  Arms: experimental
Drug: corticosteroid injection — Under sterile conditions, patients will receive a 5cc injection consisting of 2cc 1% lidocaine, 2cc 0.5% ropivacaine, and 1cc kenalog corticosteroid (40mg/cc) into the subacromial space utilizing a posterior lateral approach. Patients will be observed for 10 min in clinic for any adverse reactions.
  Other Names: triamcinalone; naropin; xylocaine
  Arms: control

SUMMARY:
The purpose of this investigator initiated study is to clinically evaluate the efficacy of a new treatment for subacromial impingement syndrome and partial thickness rotator cuff tears. This treatment consists of a platelet rich plasma injection into and around the rotator cuff. It is thought that this treatment will dramatically improve outcomes for patients suffering from these two conditions.

Subjects will be randomized by choosing a slip of paper from an envelope. This process will randomize 25 patients to the experimental group, and 25 patients to the control. The experimental group will undergo a blood draw, allowing for an injection of platelet rich plasma around the rotator cuff. The control group will undergo a corticosteroid injection into the subacromial space surrounding the rotator cuff as sole treatment. Patients will be followed for three months for pain, and will fill out questionnaires at six weeks and three months post injection, which will give insight into functionality and pain changes that the rotator cuff is experiencing due to treatment.

Subjects will be outpatients. Subjects may include employees, students, minorities, and elderly, although no subsets of these will be formed.

Subjects will be between 18 and 89 years of age.

In total, subject participation will last approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with rotator cuff symptoms for at least 4 weeks
2. Examination reveals diffuse pain with provocative maneuvers
3. Impingement symptoms with or without a partial thickness tear (if available MRI study must be less than 50% tear)
4. Willingness to participate in an investigational technique
5. Willingness to forgo any other concomitant conservative treatment modality including NSAID (must be stopped for at least one week)

Exclusion Criteria:

1. Previous rotator cuff repair
2. Complete rotator cuff tear or two tendon tears
3. Pt w/ complex regional pain syndrome
4. Cervical neuropathy or other nerve pathology
5. RA, local or systemic infection, PVD, metabolic disease such as gout, clotting disorder, anticoagulation therapy
6. Evidence of intraarticular arthritis
7. Work related or compensable injury
8. Previous treatment: corticosteroid injection in the last 6 months
9. Patients who are currently pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Montri D Wongworawat, MD, Principal Investigator — Loma Linda University Department of Orthopedics
Locations (1):
- Loma Linda University, Loma Linda, California, United States

REFERENCES:
- [Background] Fukuda H. The management of partial-thickness tears of the rotator cuff. J Bone Joint Surg Br. 2003 Jan;85(1):3-11. doi: 10.1302/0301-620x.85b1.13846. No abstract available. PMID 12585570
- [Background] Blair B, Rokito AS, Cuomo F, Jarolem K, Zuckerman JD. Efficacy of injections of corticosteroids for subacromial impingement syndrome. J Bone Joint Surg Am. 1996 Nov;78(11):1685-9. doi: 10.2106/00004623-199611000-00007. PMID 8934482
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Buchbinder R, Green S, Youd JM. Corticosteroid injections for shoulder pain. Cochrane Database Syst Rev. 2003;2003(1):CD004016. doi: 10.1002/14651858.CD004016. PMID 12535501

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: corticosteroid injection into subacromial space
  corticosteroid injection : Under sterile conditions, patients will receive a 5cc injection consisting of 2cc 1% lidocaine, 2cc 0.5% ropivacaine, and 1cc kenalog corticosteroid (40mg/cc) into the subacromial space utilizing a posterior lateral approach. Patients will be observed for 10 min in clinic for any adverse reactions.
- Experimental: patients will receive an injection of platelet rich plasma into the subacromial space
  platelet rich plasma injection : 45 ml of a patient's own blood will be collected via blood draw, maintaining sterile technique. This will then be spun down using a Magellan Autologous Platelet Separator System, yielding platelet rich plasma (PRP). Under sterile conditions, patients will receive a 5 cc PRP injection (consisting of their own PRP) with 1 cc of 1% lidocaine and 1 cc of 0.5% ropivacaine into the subacromial space, administered by an orthopedic surgeon. This will be done using a posterior lateral approach. The patient will be monitored for 10 minutes in clinic for adverse reactions.
Period: Overall Study
Arm/Group | Control | Experimental
Started | 5 | 7
Completed | 2 | 6
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (6.4) | 59.3 (14.7) | 59.25 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Pain and Disability of the Shoulder Through Validated Questionnaires
Description: Patients will be asked to fill out questionnaires to provide insight into how their condition is progressing, consisting of components of the American Shoulder and Elbow Surgeons (ASES) total score. The maximum score is 100, made up by pain and function components' sums. Only the total score is recorded, 100 being full normal function without pain, 0 being severe pain and no function.
Time Frame: 6 weeks from initial injection of corticosteroid versus platelet rich plasma
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 2 | 6
units on a scale | 81.6 (9.4) | 70.0 (13.7)

2. Primary Outcome: Pain and Disability of the Shoulder Through Validated Questionnaires
Description: as for outcome 1
Time Frame: 12 weeks from initial injection of corticosteroid versus platelet rich plasma
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 2 | 6
units on a scale | 41.6 (4.7) | 86.1 (17.1)

3. Primary Outcome: Pain and Disability of the Shoulder Through Validated Questionnaires
Description: as for outcome 1
Time Frame: 15 minutes prior to initial injection of corticosteroid versus platelet rich plasma
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 2 | 6
units on a scale | 35.0 (18.9) | 43.9 (7.4)

ADVERSE EVENTS:
Arm/Group | Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes